CLINICAL TRIAL: NCT02458027
Title: Acute Food INtake Effect of Hemp Protein (A FINEH Protein) Trial - Part 2 - Are Acute Effects of Hemp Protein on Blood Glucose and Appetite Insulin-dependent?
Brief Title: Acute Food INtake Effect of Hemp Protein (A FINEH Protein) Trial - Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Harvest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B2014:115-3
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Prevention; Obesity Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- 20g Hemp Protein Shake (Experimental): Hemp protein shake, 20 grams, given once at beginning of acute trial.
  Interventions: Dietary Supplement: Hemp Shake
- 40 g Hemp Protein (Experimental): Hemp protein shake, 40 grams, given once, at beginning of acute trial.
  Interventions: Dietary Supplement: Hemp
- 20 g Soybean Protein Shake (Active Comparator): Soybean protein shake, 20 grams, given once, at beginning of acute trial.
  Interventions: Dietary Supplement: Soybean Shake
- 40 g Soybean Protein (Experimental): Soybean protein shake, 40 grams, given once, at beginning of acute trial.
  Interventions: Dietary Supplement: Soybean
- Control Shake (Placebo Comparator): Non-protein control shake, given once, at beginning of acute trial.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Hemp Shake — Hemp Protein
  Arms: 20g Hemp Protein Shake
Dietary Supplement: Hemp — Hemp Protein Shake
  Arms: 40 g Hemp Protein
Dietary Supplement: Soybean Shake — Soybean Protein
  Arms: 20 g Soybean Protein Shake
Dietary Supplement: Soybean — Soybean Protein Shake
  Arms: 40 g Soybean Protein
Dietary Supplement: Control — Non-Protein Shake
  Arms: Control Shake

SUMMARY:
The objectives of this trial are to investigate whether the effects of hemp protein on glycemic and appetite control are insulin-dependent by measuring 1) blood glucose, insulin and appetite for one hour following consumption, 2) blood glucose, insulin and appetite following a fixed energy meal to determine the "second meal effect" of hemp protein versus soybean protein and a non-protein control.

DETAILED DESCRIPTION:
The objectives of this trial are to investigate whether the effects of hemp protein on glycemic and appetite control are insulin-dependent by measuring 1) blood glucose, insulin and appetite for one hour following consumption, 2) blood glucose, insulin and appetite following a fixed energy meal to determine the "second meal effect" of hemp protein versus soybean protein and a non-protein control. The objectives of this trial are to investigate whether the effects of hemp protein on glycemic and appetite control are insulin-dependent by measuring 1) blood glucose, insulin and appetite for one hour following consumption, 2) blood glucose, insulin and appetite following a fixed energy meal to determine the "second meal effect" of hemp protein versus soybean protein and a non-protein control.

ELIGIBILITY:
Inclusion Criteria:

* Normoglycemic (<5.6 mmol/L)
* Body mass index (BMI) of 18.5-29.9 kg/m2.

Exclusion Criteria:

* Restrained eaters
* Regularly skip breakfast
* Smokers
* Those on medications that may influence study outcomes or have experienced any gastrointestinal related health conditions/surgeries over the past year.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07-13 (Actual); Study Completion 2016-07-13 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose and Insulin Concentrations | 0-200 minutes
  Measured in blood using intravenous catheter at 12 time points, used to calculate area under curve (AUC). Glucose will be determined by automated methods using Abbot Spectrum CCX Analyzer, and Insulin will be measured by commercially available RIA kits. (Composite measure)
Appetite | 0-200 minutes
  Measured by VAS Questionnaire.
Food Intake | 0-200 minutes
  Measured by fixed energy meal.
Blood Pressure | 0-200 minutes
  Measured by automated bood pressure cuff.

SECONDARY OUTCOMES:
Palatability of Treatments and Meal | 5-80 minutes
  Measured by VAS Questionnaire.
Physical Comfort | 0-200 minutes
  Measured by VAS Questionnaire.
Energy/Fatigue | 0-200 minutes
  Measured by VAS Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jones, Ph.D., Principal Investigator — University of Manitoba, Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada